CLINICAL TRIAL: NCT05951309
Title: Effect of Myoinositol on Serum Asprosin Levels in PCOS Patients
Brief Title: Myoinositol Treatment and Asprosin Levels in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Ali Cenk, Associate Professor, Cyprus International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Asprosin-PCOS
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: PCOS; Insulin Resistance
Keywords: Polycystic ovary syndrome; Myoinositol; Metformin; Insulin resistance; Asprosin
MeSH Terms: conditions — Insulin Resistance; Polycystic Ovary Syndrome; Arachnodactyly | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myoinositol+D-chiroinositol+folic acid group (Experimental): This group is given myoinositol+d-chiro inositol+folic acid once a day (inofolic combi, ITF company, Italy) (myoinositol 550 miligram+ d-chiroinositol 13,8 miligram+folic acid 200 micrograms)
  Interventions: Drug: inofolic combi
- Metformin group (Experimental): This group is given metformin 500 miligram three times a day (glucophage 500mg, Merck company, Turkey) (total dose of metformin 1500 miligram a day)
  Interventions: Drug: Glucophage 500Mg Tablet

INTERVENTIONS:
Drug: inofolic combi — The patients in this group were given inofolic combi once a day for 12-16 weeks
  Other Names: inofolic combi, ITF company
  Arms: Myoinositol+D-chiroinositol+folic acid group
Drug: Glucophage 500Mg Tablet — The patients in this group were given glucophage three times a day for 12-16 weeks
  Other Names: glucophage, Merck company
  Arms: Metformin group

SUMMARY:
Policystic ovary syndrome is the most common endocrinopthy during reproductive period. One of the factors implicated in the pathogenesis is insulin resistance. Asprosin, which is secreted from white adipose tissue is a new candidate for insulin resistance. Myoinositol is known to reduce insulin resistance in PCOS patients. The effect of myoinsitol on serum asprosin levels is unknown yet. This study aimed to evaluate the effect of myoinositol on serum asprosin levels in PCOS patients.

DETAILED DESCRIPTION:
In addition to being the most common reproductive endocrinopathy in the population, polycystic ovary syndrome (PCOS) also carries a significantly increased risk for metabolic syndrome and type 2 diabetes. Insulin resistance and hyperinsulinemia are common findings in women with PCOS and are among the most contributing factors to hyperandrogenism in PCOS. This situation directly increases both ovarian and adrenal androgen release.

Because of the pathophysiological link between insulin resistance and PCOS, insulin sensitizers have been used in treatment of the disease through this mechanism. Metformin is the most common insulin sensitizer used in many countries for type 2 diabetes and non-diabetic patients with high insulin resistance with PCOS in the last 50 years. Current evidence suggests that metformin may have metabolic and reproductive system benefits, such as weight loss, insulin resistance, and reduction of androgen levels, as well as restoration of normal menstrual cycle and ovulation. However, major side effects such as nausea, vomiting, and gastrointestinal discomfort limit metformin use. The poor compliance observed with metformin use has prompted clinicians worldwide to find new approaches for PCOS.

Myo-inositol (MI) and d-chiro-inositol (DCI) are two of the 9 isomers of vitamin B6. MI and DCI, a naturally occurring compound, has been increasingly investigated over the past decade for its insulin sensitizing effects. As the postreceptor second messenger of the insulin signal, it interacts with GLUT4 via membrane-bound sodium-dependent channels and reduces hyperinsulinemia. Also, MI improves ovarian function, decreases lutinizing hormone / follicle stimulating hormone (LH / FSH) ratio, serum androgens, total testosterone and free testosterone levels.

Asprosin is a newly discovered peptide hormone associated with insulin resistance and increases hepatic glucose production. Produced from abnormally increased white adipose tissue in insulin resistant mammals. A recent study found that serum asprosin levels were elevated in PCOS patients and this was positively correlated with insulin resistance.

Based on these data, it has been suggested that the known positive effects of MI + DCI (inofolic combi) and metformin treatments on insulin resistance may also be on serum asprosin levels. This effect will be demonstrated with this study.

In this study, it was aimed to investigate and to compare the change on serum asprosin levels in patients with polycystic ovary syndrome after the treatment with metformin or myo-inositol + d-chiro inositol + folic acid.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome patients between 18-40 ages

Exclusion Criteria:

* Tiroid disease
* Cardiovascular disease
* Diabetes mellitus
* Smoking
* Using insulin sensitizing drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-06-03 (Actual)

PRIMARY OUTCOMES:
Serum asprosin levels 1 | Second or third day of menstruation
  First measurement of serum asprosin level at initial examination
Serum asprosin levels 2 | After 12-16 weeks from first examination
  Serum asprosin levels after 12-16 weeks from initial examination

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University Faculty of Medicine, Nicosia, Cyprus

REFERENCES:
- [Background] Diamanti-Kandarakis E, Dunaif A. Insulin resistance and the polycystic ovary syndrome revisited: an update on mechanisms and implications. Endocr Rev. 2012 Dec;33(6):981-1030. doi: 10.1210/er.2011-1034. Epub 2012 Oct 12. PMID 23065822
- [Background] Goodarzi MO, Korenman SG. The importance of insulin resistance in polycystic ovary syndrome. Fertil Steril. 2003 Aug;80(2):255-8. doi: 10.1016/s0015-0282(03)00734-9. No abstract available. PMID 12909480
- [Background] Kirpichnikov D, McFarlane SI, Sowers JR. Metformin: an update. Ann Intern Med. 2002 Jul 2;137(1):25-33. doi: 10.7326/0003-4819-137-1-200207020-00009. PMID 12093242
- [Background] Bargiota A, Diamanti-Kandarakis E. The effects of old, new and emerging medicines on metabolic aberrations in PCOS. Ther Adv Endocrinol Metab. 2012 Feb;3(1):27-47. doi: 10.1177/2042018812437355. PMID 23148192
- [Background] Palomba S, Falbo A, Zullo F, Orio F Jr. Evidence-based and potential benefits of metformin in the polycystic ovary syndrome: a comprehensive review. Endocr Rev. 2009 Feb;30(1):1-50. doi: 10.1210/er.2008-0030. Epub 2008 Dec 4. PMID 19056992
- [Background] Fulghesu AM, Romualdi D, Di Florio C, Sanna S, Tagliaferri V, Gambineri A, Tomassoni F, Minerba L, Pasquali R, Lanzone A. Is there a dose-response relationship of metformin treatment in patients with polycystic ovary syndrome? Results from a multicentric study. Hum Reprod. 2012 Oct;27(10):3057-66. doi: 10.1093/humrep/des262. Epub 2012 Jul 10. PMID 22786777
- [Background] Carlomagno G, Unfer V. Inositol safety: clinical evidences. Eur Rev Med Pharmacol Sci. 2011 Aug;15(8):931-6. PMID 21845803
- [Background] Ozay AC, Emekci Ozay O, Okyay RE, Cagliyan E, Kume T, Gulekli B. Different Effects of Myoinositol plus Folic Acid versus Combined Oral Treatment on Androgen Levels in PCOS Women. Int J Endocrinol. 2016;2016:3206872. doi: 10.1155/2016/3206872. Epub 2016 Nov 2. PMID 27882049
- [Background] Emekci Ozay O, Ozay AC, Cagliyan E, Okyay RE, Gulekli B. Myo-inositol administration positively effects ovulation induction and intrauterine insemination in patients with polycystic ovary syndrome: a prospective, controlled, randomized trial. Gynecol Endocrinol. 2017 Jul;33(7):524-528. doi: 10.1080/09513590.2017.1296127. Epub 2017 Mar 3. PMID 28277112
- [Background] Li X, Liao M, Shen R, Zhang L, Hu H, Wu J, Wang X, Qu H, Guo S, Long M, Zheng H. Plasma Asprosin Levels Are Associated with Glucose Metabolism, Lipid, and Sex Hormone Profiles in Females with Metabolic-Related Diseases. Mediators Inflamm. 2018 Nov 6;2018:7375294. doi: 10.1155/2018/7375294. eCollection 2018. PMID 30524197
- [Background] Alan M, Gurlek B, Yilmaz A, Aksit M, Aslanipour B, Gulhan I, Mehmet C, Taner CE. Asprosin: a novel peptide hormone related to insulin resistance in women with polycystic ovary syndrome. Gynecol Endocrinol. 2019 Mar;35(3):220-223. doi: 10.1080/09513590.2018.1512967. Epub 2018 Oct 16. PMID 30325247